CLINICAL TRIAL: NCT03346460
Title: Effect of Photodymamic Therapy With Urucum and LED in the Reduction of Halitosis: a Clinical and Microbiological Trial
Brief Title: Effect of Photodymamic Therapy With Urucum and LED in the Reduction of Halitosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Marcela Leticia Leal Gonçalves, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALIURU
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tongue scraper group (Group 1) (Experimental): Fifteen patients will be included in this group. Tongue scraping will be performed by the same operator in all patients. Posterior-anterior movements will be performed with the scraper over the lingual dorsum, followed by cleaning the scraper with a gauze. This procedure will be performed ten times in each patient, in order to standardize the mechanical removal of the tongue coating.
  Interventions: Other: Tongue Scraping
- aPDT group (Group 2) (Experimental): Fifteen patients will be included in this group. One session of aPDT will be performed with the photosensitizer (PS) urucum manipulated at a concentration of 20% (Fórmula e Ação®) in spray, to be applied in sufficient quantity to cover the middle third and back of the tongue (5 sprinkles) for 5 minutes for incubation. The excess will be removed with a sucker in order to keep the surface wet with the PS itself, without using water. Six points with a distance of 1 cm between them will be irradiated, considering the halo of light scattering and effectiveness of aPDT. The apparatus shall be precalibrated at wavelength 440-480nm for 60 seconds per point, irradiance of 450mW/cm and the light shall be irradiated so that a halo of 2cm diameter is formed per point.
  Interventions: Radiation: aPDT
- Tongue scraper and aPDT (Group 3) (Experimental): Tongue scraping will be performed by the same operator in all patients. Posterior-anterior movements will be performed with the scraper over the lingual dorsum, followed by cleaning the scraper with a gauze. This procedure will be performed ten times in each patient, in order to standardize the mechanical removal of the tongue coating. After, one session of aPDT will be performed with the photosensitizer (PS) urucum manipulated at a concentration of 20% (Fórmula e Ação®) in spray, to be applied in sufficient quantity to cover the middle third and back of the tongue (5 sprinkles) for 5 minutes for incubation. Six points with a distance of 1 cm between them will be irradiated, considering the halo of light scattering and effectiveness of aPDT. The apparatus shall be precalibrated at wavelength 440-480nm for 60 seconds per point, irradiance of 450mW/cm and the light shall be irradiated so that a halo of 2cm diameter is formed per point.
  Interventions: Radiation: Tongue scraper and aPDT

INTERVENTIONS:
Other: Tongue Scraping — Tongue scraping will be performed by the same operator in all patients. Posterior-anterior movements will be performed with the scraper over the lingual dorsum, followed by cleaning the scraper with a gauze. This procedure will be performed ten times in each patient, in order to standardize the mechanical removal of the tongue coating.
  Arms: Tongue scraper group (Group 1)
Radiation: aPDT — One session of aPDT will be performed with the photosensitizer (PS) urucum manipulated at a concentration of 20% (Fórmula e Ação®) in spray, to be applied in sufficient quantity to cover the middle third and back of the tongue (5 sprinkles) for 5 minutes for incubation. The excess will be removed with a sucker in order to keep the surface wet with the PS itself, without using water. Six points with a distance of 1 cm between them will be irradiated, considering the halo of light scattering and effectiveness of aPDT. The apparatus shall be precalibrated at wavelength 440-480nm for 60 seconds per point, irradiance of 450mW/cm and the light shall be irradiated so that a halo of 2cm diameter is formed per point.
  Arms: aPDT group (Group 2)
Radiation: Tongue scraper and aPDT — Tongue scraping will be performed by the same operator in all patients. Posterior-anterior movements will be performed with the scraper over the lingual dorsum, followed by cleaning the scraper with a gauze. This procedure will be performed ten times in each patient, in order to standardize the mechanical removal of the tongue coating. After, one session of aPDT will be performed with the photosensitizer (PS) urucum manipulated at a concentration of 20% (Fórmula e Ação®) in spray, to be applied in sufficient quantity to cover the middle third and back of the tongue (5 sprinkles) for 5 minutes for incubation. Six points with a distance of 1 cm between them will be irradiated, considering the halo of light scattering and effectiveness of aPDT. The apparatus shall be precalibrated at wavelength 440-480nm for 60 seconds per point, irradiance of 450mW/cm and the light shall be irradiated so that a halo of 2cm diameter is formed per point.
  Arms: Tongue scraper and aPDT (Group 3)

SUMMARY:
Halitosis, also known as bad breath, is a term used to define an unpleasant and foul odor that emanates from the mouth and may have local or systemic origin. This project aims to observe the presence of halitosis and to verify if the treatment with antimicrobial photodynamic therapy (aPDT) is effective against it. The investigators will select 45 students or UNINOVE employees, from 18 to 25 years old, with a diagnosis of halitosis, presenting sulfite (SH2) ≥ 112 ppb on gas chromatography. Patients will be randomly divided into 3 groups of 15, which will receive different treatments: Group 1: treatment with tongue scraper; Group 2: aPDT applied in the back region and middle third of the tongue; Group 3: combined treatment of tongue scraper and aPDT. For the aPDT we will use urucum manipulated in the concentration of 20% (Fórmula e Ação®) in spray, to be applied in sufficient quantity to cover the middle third and back of the tongue (5 sprinkles) for 5 minutes for incubation, associated with a LED (Valo Cordless Ultradent®). 6 points will be irradiated on the back of the tongue with a distance of 1 cm between the points, considering the halo of light scattering and effectiveness of aPDT. The apparatus shall be precalibrated at wavelength 440-480nm for 60 seconds per point, irradiance of 450mW/cm and the light shall be irradiated so that a halo of 2cm diameter is formed per point. The results of the halimetry will be compared before and immediately after the treatment, besides the microbiological analysis of the tongue coating, before and after the treatment. The normality of the data will be measured using the Shapiro-Wilk test, and in the case of normality the Variance Analysis (ANOVA) test will be applied, and in the case of non-parametric data, the Kruskal-Wallis test will be used. To analyze the results of each treatment in both periods of the study, the Wilcoxon test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years;
* Sulphide (SH2) ≥ 112 ppb in the gas chromatography.

Exclusion Criteria:

* Dentofacial anomalies (such as cleft lip and cleft palate);
* Undergoing orthodontic and/or orthopedic treatment;
* Undergoing oncological treatment;
* Systemic alterations (gastrointestinal, renal, hepatic);
* Treatment with antibiotics up to 1 month before the survey;
* Pregnant.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-12-05 (Estimated); Study Completion 2018-12-05 (Estimated)

PRIMARY OUTCOMES:
Halimetry (gas chromatography) | Through study completion, an average of 1 year.
  Oral air collection will follow the manufacturer's guidelines (Oral ChromaTM Manual Instruction) where the participant will be instructed to rinse with cysteine (10 mM) for 1 minute, then remain with his/her mouth closed for 1 minute. A syringe from the same manufacturer for collection of mouth air will be introduced into the patient's mouth. During 1 minute the patient will remain closed mouth, breathing through the nose, without touching the syringe with the tongue. The plunger will be pulled out, we will re-empty the syringe air into the patient's mouth and again pull the plunger to fill the syringe with the breath sample. We will wipe the tip of the syringe with gauze to remove moisture from the saliva, place the gas injection needle in the syringe, and adjust the plunger to 0.5 ml. The gases collected at the entrance door of the appliance are injected in a single movement. This procedure will be done before and immediately after treatment.

SECONDARY OUTCOMES:
Microbiological analysis of tongue coating | Through study completion, an average of 1 year.
  The microbiological analysis of tongue coating will be performed by collecting biofilm samples from the region of the lingual dorsum with a 1μl inoculation loop. Samples will be transferred into individual vials containing 1.5 ml of reduced transport fluid and vortexed for approximately 30 seconds. After homogenisation, the ten-fold dilution series will be prepared in 180μl sterile PBS solution and 10-2, 10-3, 10-4 and 10-5 aliquots, transferred to BHI agar plates. Considering that the main bacteria responsible for the production of CSV are Gram-negative and anaerobic, plaques will be incubated in an anaerobic jar for 72 h at 370 C, for counting of the colony-forming units (CFU) and comparison of the numbers before and immediately after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela LL Gonçalves, MS, Principal Investigator — University of Nove de Julho
Locations (1):
- UNINOVE, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Goncalves MLL, da Mota ACC, Deana AM, Guedes GH, Cavalcante LAS, Prates RA, Horliana ACRT, Pavani C, Motta LJ, Bitencourt GB, Fernandes KPS, Salgueiro MDCC, Mesquita-Ferrari RA, da Silva DFT, Franca CM, Bussadori SK. Photodynamic therapy with Bixa orellana extract and LED for the reduction of halitosis: study protocol for a randomized, microbiological and clinical trial. Trials. 2018 Oct 29;19(1):590. doi: 10.1186/s13063-018-2913-z. PMID 30373650